CLINICAL TRIAL: NCT06597149
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on Plasma Insulin Levels
Acronym: TaVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Principal Investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24300
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Healthy; Individual

STUDY DESIGN:
Intervention Model Description: Healthy adults will receive mild transcutaneous stimulation of the auricular branch of the vagal nerve in order to determine if the stimulation affects plasma insulin levels.
Masking Description: Individuals will be either assigned to either the Active or the Sham groupings. The active group will receive a mild stimulation from the TaVNS device and the sham group will receive no stimulation but will believe that they are receiving a stimulus.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Stimulation (Experimental): Subjects are placed supine, ECG electrodes are applied, a butterfly catheter is inserted into a peripheral vein. A 5 ml sample of blood is withdrawn. A TENS device is placed on the cutaneous branch of the auricular branch of the vagus nerve. After a twenty-minute baseline reading, the TENS unit is then turned ON and electrical stimuli are delivered over 40 minutes. A second sample of blood representing the experimental period is drawn at the end of the 40 minutes. The TENS device is then turned to the OFF positon and after twenty minutes a third and final sample of blood is drawn.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Healthy adult participants will be assigned to either the stimulation group or the sham group. The stimulation group will receive mild stimulation from the TeNS device and the sham group will receive no stimulation but will believe that they are receiving stimulus.

SUMMARY:
The purpose of this study is to find out if investigators can stimulate the vagus nerve (a nerve in the body that runs from your brain to the large intestine), and influence insulin, C-peptide, and glucose levels. C-peptide is a substance that is created when insulin is produced and released into the body. The vagus nerve is a largely internal nerve that controls many bodily functions, including stomach function.

Investigators hope that by stimulating the vagal nerve using the TeNS behind the ear, this stimulation can affect insulin levels, and this will help innovate treatment of patients with nausea, vomiting, and disordered stomach function, and patients with diabetes.

Researchers hope to be able to measure the activity of the vagus nerve when it is stimulated in other ways. This could help investigators learn more about studying this nerve in the future.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary: The research described in this protocol is best described as an extension of the researcher's current protocol which is designed to measure cervical compound vagal nerve action potentials in patients who have an implanted gastric electrical stimulation device (GESD). The difference is that only healthy volunteer subjects will be recruited and studied, and rather than undergoing gastric electrical stimulation (GES), volunteer subjects will undergo transcutaneous stimulation of the auricular branch of the vagus nerve (taVNS) to determine whether this modality will also influence plasma insulin, C-peptide and glucose levels. While not a part of the current proposal; if the results of this study are promising we anticipate applying electrical stimulation of the ABVN in future studies of gastroparetic patients with symptomatic nausea and vomiting.

Secondary/exploratory: If taVNS proves to have an effect on circulating plasma insulin levels, then a secondary component of this study is to determine which subject variables (age, gender, BMI) may influence this response. While not formally a part of this proposal, investigators anticipate future studies will be designed to determine the optimal stimulus parameters (stimulus current, frequency, pulse duration) needed to produce this effect. Researchers' previous investigation using percutaneous electrical nerve field stimulation (PENFS) have shown that this modality affects the sympathetic and parasympathetic controls or heart rate variability. The current proposal will also determine whether the same effect occurs with transcutaneous auricular vagus nerve stimulation (taVNS).

SPECIFIC AIM 1:

To determine if acute taVNS stimulation of the cymba concha area of the external ear in human subjects affects plasma insulin, C-peptide, and glucose levels.

Investigators' preliminary studies show that electrical stimuli applied to electrodes implanted in the serosa of the stomach augment plasma insulin levels in humans. Presumably this is due activation of sympathetic and parasympathetic nerves which also innervate the pancreas. Researchers propose to non-invasively access the vagus nerve by applying electrical stimuli to the cymba concha area of the human external ear. This area is innervated by the cutaneous branch of the vagus nerve which, in turn, sends branches to the sensory nucleus of the vagus nerve, the nucleus tractus solitarius, which then sends nerve fibers throughout the brainstem to control autonomic function throughout the autonomic nervous system.

SPECIFIC AIM 2:

To determine if acute taVNS of the cymba concha area of the external ear affects heart rate variability in human subjects.

Heart rate variability is governed by parasympathetic and sympathetic nerves. By using frequency-domain and time domain analysis it is possible to determine whether 1) taVNS activates the auricular branch of the vagus nerve, and 2) whether any observed effects are mediated through the parasympathetic and/or sympathetic autonomic nervous system.

SPECIFIC AIM 3:

To determine if the changes in plasma insulin, C-peptide, or glucose levels are associated with corresponding changes in parasympathetic or sympathetic activation.

By using frequency-domain and time-domain analysis of heart rate variability it is possible to determine whether any observed changes are due to activation of parasympathetic or sympathetic nervous system or a combination of both. Some subjects may show a greater change in plasma insulin, C-peptide or glucose levels than others during taVNS. Researchers propose to determine whether these changes are mirrored by corresponding alterations in parasympathetic and sympathetic nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Aged 18-70
* Willing to have ECG electrodes placed on their neck and chest areas.
* Willing to have electrodes placed in the external ear.
* Willing to have an indwelling catheter placed to avoid multiple sticks for blood draw.

Exclusion Criteria:

* Unable to provide consent.
* Diabetes diagnosis per patient report
* Having known allergies to adhesive on electrode pads or bandages
* Having gastric motility issues as determined by the PI or clinical coordinator.
* Taking any medications that may affect gastric motility or cardiac variability, i.e. alpha or beta blockers for hypertension.
* Pregnant females
* Those unwilling to have the taVNS device placed in their ear.
* Those unwilling to consent to a blood draw.
* Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Association between acute transcutaneous auricular vagus nerve stimulation and change in plasma insulin levels | one month
  Repeated measures analysis of variance will be used to determine the effects of stimulation period (baseline, end of stimulation, end of non-stimulation) and active/control group on plasma insulin levels.
Association between acute transcutaneous auricular vagus nerve stimulation and change in C-peptide levels | one month
  - Measure description: Repeated measures analysis of variance will be used to determine the effects of stimulation period (baseline, end of stimulation, end of non-stimulation) and active/control group on C-peptide levels.
Association between acute transcutaneous auricular vagus nerve stimulation and change in glucose levels | one month
  Repeated measures analysis of variance will be used to determine the effects of stimulation period (baseline, end of stimulation, end of non-stimulation) and active/control group on glucose levels
Association between acute transcutaneous auricular vagus nerve stimulation and heart rate variability | one month
  Repeated measures analysis of variance will be used to determine the effects of stimulation period (baseline, end of stimulation, end of non-stimulation) and active/control group on heart rate variability.
Association between changes in heart rate variability and plasma insulin levels | one month
  Pearson's correlation coefficients will be used to evaluate the association between change in heart rate variability (end of stimulation minus baseline) with changes in plasma insulin levels (end of stimulation minus baseline). Heart rate variability will be used as an indication of changes in parasympathetic or sympathetic activation.
Association between changes in heart rate variability and C-peptide levels | one month
  Pearson's correlation coefficients will be used to evaluate the association between change in heart rate variability (end of stimulation minus baseline) with changes in C-peptide levels (end of stimulation minus baseline). Heart rate variability will be used as an indication of changes in parasympathetic or sympathetic activation.
Association between changes in heart rate variability and glucose levels | one month
  Pearson's correlation coefficients will be used to evaluate the association between change in heart rate variability (end of stimulation minus baseline) with changes in glucose levels (end of stimulation minus baseline). Heart rate variability will be used as an indication of changes in parasympathetic or sympathetic activation.

SECONDARY OUTCOMES:
Correlation between gender and changes in circulating plasma insulin levels | one month
  Pearson's correlation coefficient will be calculated for the association between change in circulating plasma insulin levels (end of stimulation minus baseline) and patient gender.
Correlation between age and changes in circulating plasma insulin levels | one month
  Pearson's correlation coefficient will be calculated for the association between change in circulating plasma insulin levels (end of stimulation minus baseline) and patient age.
Correlation between body mass index and changes in circulating plasma insulin levels | one month
  Pearson's correlation coefficient will be calculated for the association between change in circulating plasma insulin levels (end of stimulation minus baseline) and patient body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Nowak, MD, Principal Investigator — IU Medical Scool
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
The blood samples collected will be processed in the CRC lab to obtain blood serum. This serum will then be transferred to Dr. Robert Considine at the Indiana University Center for Diabetes and Metabolic Diseases. These samples will only be identified with the study subject number and which blood draw number (1,2,3) the vial contains.
  ECG recordings are digitized and downloaded to a computer and are analyzed using heart rate variability software (LABVIEW, AD Instruments, Boston, MA). This software contains no references to any person and only contains the subject number for the study.

REFERENCES:
- [Background] van der Voort IR, Becker JC, Dietl KH, Konturek JW, Domschke W, Pohle T. Gastric electrical stimulation results in improved metabolic control in diabetic patients suffering from gastroparesis. Exp Clin Endocrinol Diabetes. 2005 Jan;113(1):38-42. doi: 10.1055/s-2004-830525. PMID 15662594
- [Background] Huang F, Dong J, Kong J, Wang H, Meng H, Spaeth RB, Camhi S, Liao X, Li X, Zhai X, Li S, Zhu B, Rong P. Effect of transcutaneous auricular vagus nerve stimulation on impaired glucose tolerance: a pilot randomized study. BMC Complement Altern Med. 2014 Jun 26;14:203. doi: 10.1186/1472-6882-14-203. PMID 24968966
- [Background] Vosseler A, Zhao D, Fritsche L, Lehmann R, Kantartzis K, Small DM, Peter A, Haring HU, Birkenfeld AL, Fritsche A, Wagner R, Preissl H, Kullmann S, Heni M. No modulation of postprandial metabolism by transcutaneous auricular vagus nerve stimulation: a cross-over study in 15 healthy men. Sci Rep. 2020 Nov 24;10(1):20466. doi: 10.1038/s41598-020-77430-2. PMID 33235256
- [Background] Kozorosky EM, Lee CH, Lee JG, Nunez Martinez V, Padayachee LE, Stauss HM. Transcutaneous auricular vagus nerve stimulation augments postprandial inhibition of ghrelin. Physiol Rep. 2022 Apr;10(8):e15253. doi: 10.14814/phy2.15253. PMID 35441808
- [Background] Yin J, Ji F, Gharibani P, Chen JD. Vagal Nerve Stimulation for Glycemic Control in a Rodent Model of Type 2 Diabetes. Obes Surg. 2019 Sep;29(9):2869-2877. doi: 10.1007/s11695-019-03901-9. PMID 31222497
- [Background] Payne SC, Ward G, Fallon JB, Hyakumura T, Prins JB, Andrikopoulos S, MacIsaac RJ, Villalobos J. Blood glucose modulation and safety of efferent vagus nerve stimulation in a type 2 diabetic rat model. Physiol Rep. 2022 Apr;10(8):e15257. doi: 10.14814/phy2.15257. PMID 35439355
- [Background] Hampton RF, Jimenez-Gonzalez M, Stanley SA. Unravelling innervation of pancreatic islets. Diabetologia. 2022 Jul;65(7):1069-1084. doi: 10.1007/s00125-022-05691-9. Epub 2022 Mar 29. PMID 35348820
- [Background] Zhu Y, Xu F, Lu D, Rong P, Cheng J, Li M, Gong Y, Sun C, Wei W, Lin L, Chen JDZ. Transcutaneous auricular vagal nerve stimulation improves functional dyspepsia by enhancing vagal efferent activity. Am J Physiol Gastrointest Liver Physiol. 2021 May 1;320(5):G700-G711. doi: 10.1152/ajpgi.00426.2020. Epub 2021 Feb 24. PMID 33624527
- [Background] Krasaelap A, Sood MR, Li BUK, Unteutsch R, Yan K, Nugent M, Simpson P, Kovacic K. Efficacy of Auricular Neurostimulation in Adolescents With Irritable Bowel Syndrome in a Randomized, Double-Blind Trial. Clin Gastroenterol Hepatol. 2020 Aug;18(9):1987-1994.e2. doi: 10.1016/j.cgh.2019.10.012. Epub 2019 Oct 14. PMID 31622740